CLINICAL TRIAL: NCT02749955
Title: Partner Services Pre-exposure Prophylaxis (PS-PrEP)
Acronym: PS-PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB14-1087
Record Dates: First submitted 2016-02-23; First posted 2016-04-25 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: HIV Transmission, Transtheoretical Model of Change
Keywords: HIV prevention; Pre exposure prophylaxis; Men who have sex with men; Partner services; Linkage to care; Seronegative; Sexually transmitted diseases
MeSH Terms: conditions — Homosexuality; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PS-PrEP Intervention Group (Experimental)
  Interventions: Behavioral: PS-PrEP Intervention Group
- PrEPLine Control Group (Active Comparator)
  Interventions: Behavioral: PrEPLine Control Group
- CDPH Prevention Projects (No Intervention)

INTERVENTIONS:
Behavioral: PS-PrEP Intervention Group — This group will involve working with a PS-PrEP social worker to learn about PrEP. The PS-PrEP social worker will help subjects develop a care plan based on the subject's decision about whether or not to use PrEP. This may include referrals for PrEP, other services, and/or HIV testing. Personal contact will continue by way of phone calls, and messages in between visits.
  Arms: PS-PrEP Intervention Group
Behavioral: PrEPLine Control Group — This group follows routine department of public health care as a Linkage to Care Specialist from the PrEPLine provides subjects with PrEP education and the ability to schedule an initial PrEP appointment. In addition to this care, subjects will be referred for additional testing for STIs/HIV and subjects will be given information about programs available to prevent HIV infection, which include PrEP.
  Arms: PrEPLine Control Group

SUMMARY:
This study evaluates the feasibility (reach, adoption, safety and implementation) and initial efficacy (higher linkage to care) of the Partner Services Pre-exposure Prophylaxis (PS-PrEP) intervention versus phone based Pre-exposure Prophylaxis (PrEP) treatment at 3 months post randomization among a sample of high risk individuals 18 - 35 years from clinic-based recruitment and internal referrals from social network based projects. The evaluation of the intervention will be used to strengthen routine department of public health services linkage to PrEP care.

DETAILED DESCRIPTION:
The investigators will enroll 150 human immunodeficiency virus (HIV) seronegative contacts presenting to sexually transmitted infections (STI) clinics for HIV testing and referrals from the Chicago Center for HIV Elimination (CCHE) network-based projects, ages 18 - 35, in this study over a period of 18 months referred from University of Chicago clinics and outreach space that perform HIV Partner Services as well as Expanded HIV testing and Linkage to Care (XTLC) and Chicago Department of Public Health (CDPH) partner notification services on the South Side of Chicago.

Eligible participants will undergo consent and complete the baseline assessment within 14 days of eligibility. Subjects will be taken through the baseline assessment includes survey modules described in detail below (demographics, substance use, mental health and stigma). At the baseline visit, the investigators will collect data on demographics and sex and drug-using risk variables. From the common electronic medical record at both clinics, the investigators will collect data on participants' care providers and health care utilization. Subjects will be asked to sign a medical release form.

Whenever possible, the investigators selected measures: (1) previously tested in HIV implementation studies, particularly among younger and minority populations and (2) to maximize comparability to other studies.

Randomization Following the baseline assessment, study participants will be randomized into one of two groups: the Partner Services Pre-exposure Prophylaxis (PS-PrEP) intervention group or the standard of care practice PrEPLine control condition. Study staff will discuss pros and cons, ethical basis of assigning participants to different arms of a study, of control and intervention with participants (equipoise induction) to balance the desirability of the two intervention conditions. Block randomization will be used for allocation to ensure balanced representation in the two treatment arms (control and intervention) as recruitment progresses. The randomization assignment will be generated using the R program. Once randomized, each participant will be given a study identification number and will be allocated to their respective study condition to begin the trial. Due to the nature of this intervention, complete masking of participants, investigators, and interventionist is not possible. The research staff will work directly with the linkage and support group. To help mitigate possible bias in interviewing, baseline data collection will occur prior to randomization.

After randomization, those who are in the intervention group will be taken through the Session I of the intervention. This may take place on the same day as the consent and baseline visit, or it may be scheduled at a different time depending the subject's availability.

2 Week Visit (Intervention Group)

The two week visit is post baseline survey and enhanced linkage to Pre-exposure Prophylaxis (PrEP) care. During the two week visit the interventionist and the participant will engage in Session II of the intervention: follow-up sessions to promote PrEP linkage and retention. During this session, the interventionist will check-in with participant in-person or telephonically. This follow-up visit will be integrated into Components 2 & 3 of the intervention, mini-booster sessions and best linkage practices, as described below.

3 Month Visit

During the three-month visit the control and the intervention arms will come in to take their survey. The survey is composed entirely of survey instruments taken from the baseline survey, including those that capture attitudes towards PrEP, HIV, risk behaviors, and self-perception of risk. This survey will allow the research staff to track changes over time with intermittent assessments.

6 Month Visit (Intervention Group)

Participants in the intervention arm will be contacted after six months for a scheduled mini-booster session. At that time, those participants who report significant barriers to PrEP adherence, or who express a desire to engage (or re-engage) in linkage to PrEP care will be scheduled for an additional in-person intervention session. The purpose of this follow-up sessions is to assess (and re-assess) the success of the linkage to PrEP care, to address barriers to PrEP adherence, and to refine participants' "linkage roadmap" to support future PrEP adherence.

12 Month Visit

During the twelve month visit the control and the intervention arms will come in to take their survey. The survey is composed entirely of survey instruments taken from the baseline survey, including those that capture attitudes towards PrEP, HIV, risk behaviors, and self-perception of risk. This survey will allow the research staff to track changes over time with intermittent assessments.

Linkage and Support Group

Component 1 Face to face intervention Session 1

The first and main component of the PS-PrEP intervention consists of an intervention session with the study participant which takes approximately 65 minutes. The structure and content of the face to face session is theoretically and empirically grounded, and review four primary content areas: (1) to provide information on PrEP and an overview of the linkage to care process; (2) to introduce participants to the cognitive-behavioral therapy (CBT) framework; (3) to use Motivational Interviewing techniques to build upon participants' motivation to reduce their HIV risk; and (4) to develop a plan to address barriers to PrEP linkage through the development of a Linkage Roadmap.

The conceptual framework guiding this session is the Information Motivation Behavior (IMB) model, designed to target the client's knowledge, personal and social motivation to engage in linkage, and their self-efficacy and objective ability (i.e., behavioral skills) to follow through with linkage to PrEP care. In addition, the session also provides clients with the knowledge and skills necessary to target their motivational readiness (i.e., their stage of change), expectancies and self-efficacy to get linked to care, thus, targeting determinants of linkage to care.

The first area is informational and reviews PrEP in general and linkage to PrEP care. PrEP knowledge is adapted from the Center for Disease Control (CDC) training modules that are part of the Sustainable Health Center Implementation PrEP Pilot (SHIPP) project. Linkage best practices are based upon linkage to HIV care and our current practices within the University of Chicago, XTLC and the CDPH linkage to care working group.

The second area is based on the CBT framework that focuses on examining one's relationship between thoughts, feelings, and behaviors. CBT has been shown to be an effective intervention technique to improve both psychosocial outcomes as well as medical adherence in a variety of settings.

The third area of Motivational Interviewing focuses on motivational processes that facilitate change within an individual Motivational Interviewing is a fundamentally client-centered and collaborative clinical approach, which honors patients' autonomy and is guided by patients' own intrinsic motivation for change.

Finally, the fourth component of this session, the Linkage Roadmap, is adapted from the intervention research of Safren et al. and utilizes CBT techniques to promote health and medication adherence among people living with HIV/AIDS. Through the vehicle of the Linkage Roadmap, the client and interventionist will collaboratively develop an individualized PrEP linkage, adherence, and retention plan. In the process, the interventionist will lead the client through a problem-solving activity to identify and address anticipated barriers to PrEP linkage. This interactive activity targets the behavioral skills component of IMB and the expectancies and self-efficacy, and has been utilized in a wide range of HIV/AIDS-related interventions.

Component 2 (Weeks 1-12) Mini-Booster Sessions

The booster sessions, as outlined in the final section of the Intervention Manual, will be conducted by the using a method selected by the subject which can include a by phone call, text messaging, or private message through social networking such as Facebook and will be relatively short in duration (5-6 minutes). This second component will be completed in tandem with component 3 below. The primary purposes of the boosters are to "check-in" with the client about their experience getting linked to care, to answer any questions they may have with respect to the, to review the Linkage Roadmap, and to problem solve with them if they have been experiencing any difficulties enacting the Linkage Roadmap. The structured content of each booster session will map directly onto a component of the face to face intervention session that lasted for 25 minutes (therefore four 5-6 minute structural content components). In our experience, a combination of synchronous and asynchronous communication has been effective in piloting the mini-boosters. A large body of research indicates that brief telephonic booster sessions (synchronous communication) offered as supplemental support to multi-component interventions similar to the proposed PS-PrEP protocol are associated with increased and sustained behavior change. The idea is to keep intervention content and form salient and to provide the participant with individualized support to utilize the skills and information imparted during the face-to-face intervention. In total, the investigators will deliver 4 booster sessions. The first two booster sessions will occur once every week for the first two weeks and the second two boosters monthly thereafter. Booster sessions will continue until the client has either been linked to care (completed 2 clinic visits) or the three month linkage to care window has closed. The flexibility of the booster sessions are designed to tailor the intervention to participants who may need a higher level of support to adhere to the Linkage Roadmap. All booster sessions will begin according to procedures to maintain confidentiality reviewed by the interventionist at baseline.

Component 3 (Weeks 1-12) Best linkage practices

Throughout the entire intervention period, research staff will engage the participant in best linkage practices, as introduced in Module C of Session I of the intervention, the "Linkage Roadmap," and incorporated into subsequent follow-up and booster sessions. This component will be conducted in tandem with component 2 above. Best linkage practices have been developed by the CDPH linkage working group have been adopted by HIV Focus. The linkage includes accompanying participants to the first and second PrEP clinical appointment. The research staff is not permitted to transport participants in their personal vehicle, however, will provide transportation vouchers as needed. The research staff will accompany participants to their first two medical appointments, unless participants state that they do not want to be accompanied. When at the clinic, the research staff will ask the participant if they would like to be accompanied when in the exam room. While waiting for the first appointment, the research staff will clearly explain the role of the clinic staff and the purpose of the additional clinic testing. The participants will be introduced to new faces and information during the first appointment. The research staff will continually clarify their role (ie. that they will not serve as participant's health care provider or case manager) and that any questions or concerns should be directed to the health care provider. During the second appointment, the research staff will help facilitate provider efforts to engage the participant, clarifying and addressing patient and provider concerns. The participant will be gently reminded during this second appointment that it will be the last appointment that the research staff will attend.

CONTROL CONDITION (Low Threshold Prevention Group)

Control condition for clients testing HIV negative through clinic-based recruitment and internal referrals includes a brief risk assessment, (which will occur prior to consenting of a subject on the study) conducted by the University of Chicago, CDPH clinic staff, and referral for additional STI testing and provision of information regarding other HIV prevention programming (including PrEP). Clients will receive low threshold intervention through the PrEP Line, a phone-based PrEP linkage intervention. The PrEPLine Linkage to Care Specialist (LTC) will establish contact with client, facilitate an initial interview to provide PrEP education, collect necessary patient information and build rapport. Once relevant information is collect, if the participant is interested and eligible for PrEP, LTC specialist will collaboratively determine most appropriate PrEP provider (based on location, insurance, and patient preference) and will offer to schedule initial PrEP appointment.

Once clients engage in PrEP care, routine care is comprehensive and is adapted from the CDC's and Fenway Institute's interim guidance for clinicians considering the use of PrEP (with an update for injecting drug users).

The University of Chicago faculty clinicians at both clinical PrEP sites, University of Chicago and Access Grand Boulevard, also provide HIV primary care services and include mental health services and psychosocial support services. The initial visit of an eligible PrEP client is primarily to receive information on PrEP and undergo an initial medical assessment, usually with follow-up 2 weeks later. In contrast to Ryan White HIV/AIDS Programming for HIV infected clients, there is no formal intake visit with case management follow-up which affords a much more streamlined process for care provision.

The referral to STI testing and HIV prevention programming (including PrEP) by disease intervention specialist staff, potential visits with PrEP care providers including any required mental health services that occur during the first 2 weeks and then at 3 month intervals thereafter constitute treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* HIV seronegative and completed post-test counseling
* Eligible for PrEP according to the package insert
* 18 - 35 years of age
* African American/Black identified MSM
* English speaking
* Owns a cell phone not shared with other persons
* Agreeable to text/phone mini-booster sessions; and
* Lives in the Chicago metropolitan area for more than 6 months annually

Exclusion Criteria:

* Taking or taken PrEP in the previous 12 months
* Unable to provide consent
* Plan to move out of the are

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Surveying the uptake of PrEP care after randomized behavioral intervention or routine linkage | One Year
  Comparing 60 individuals who receive enhanced personalized linkage to care with a social worker to 60 individuals who receive routine phone based PrEP linkage.
Timing of linkage to care after behavioral intervention | One Year
  At 6 and 12 months linkage to care will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Teixeira da Silva D, Bouris A, Ramachandran A, Blocker O, Davis B, Harris J, Pyra M, Rusie LK, Brewer R, Pagkas-Bather J, Hotton A, Ridgway JP, McNulty M, Bhatia R, Schneider JA. Embedding a Linkage to Preexposure Prophylaxis Care Intervention in Social Network Strategy and Partner Notification Services: Results From a Pilot Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2021 Feb 1;86(2):191-199. doi: 10.1097/QAI.0000000000002548. PMID 33109935